CLINICAL TRIAL: NCT04712877
Title: LEADER Neoadjuvant Screening Trial: LCMC4 Evaluation of Actionable Drivers in Early Stage Lung Cancers
Brief Title: Testing Tumor Tissue and Blood to Help Select Personalized Treatments for Patients With Suspected Lung Cancers
Status: Recruiting | Type: Observational
Sponsor: Lung Cancer Mutation Consortium (Network)
Collaborators: Lung Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Scott J. Swanson, Canepari Family Distinguished Chair in Thoracic Surgery, Director of Minimally Invasive Thoracic Surgery and Clinical Director of Thoracic Surgery, BWH, Associate Chief of Surgery, DFCI, Professor of Surgery, Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: LCMC LEADER
Record Dates: First submitted 2020-10-16; First posted 2021-01-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ctDNA, tumor NGS — Testing for actionable oncogenic drivers
  Other Names: FoundationOne CDx; FoundationOne Liquid

SUMMARY:
This collaborative screening protocol, developed by the Lung Cancer Mutation Consortium (LCMC) and supported by the Thoracic Surgery Oncology Group (TSOG), is designed to determine the feasibility of comprehensive molecular profiling to detect actionable oncogenic drivers in patients with suspected early stage lung cancers scheduled to undergo biopsies to establish the diagnosis of lung cancer.

The primary purpose of this testing is to determine the presence of 12 oncogenic drivers (mutations in EGFR, BRAFV600E , MET exon 14, KRAS G12C and HER2, rearrangements in ALK, RET, NTRK, EGFR exon 20 insertion and ROS1, and amplification of MET and HER2) that can serve as targets making patients eligible for upcoming targeted neoadjuvant therapy trials. The ultimate goal is to use this information from the screening process to select the optimal neoadjuvant therapy and wherever possible enroll patients onto separate neoadjuvant therapy trials with genomically matched treatments or other appropriate trials if no actionable driver mutation is detected.

Thoracic Surgery Oncology Group (TSOG) is a network of surgeons within North American Thoracic Surgery Academic Centers aligned with the goal of enhancing patient care through administration of multi-site trials focused on recent advances in lung cancer. TSOG has aligned with the LCMC4 sites to enroll the LCRF-LEADER screening trial. TSOG's involvement will be essential in trial enrollment and ultimate interpretation of the multimodal clinical and translational data collected as part of this study. We estimate we will detect an actionable oncogenic driver in 33% of cases. The remaining 66% of patients will represent a cohort identified by their care teams as candidates for other potential neoadjuvant therapies which may include checkpoint inhibitors such as atezolizumab, durvalumab, nivolumab, and pembrolizumab or other novel agents.

The targeted therapy treatment trials will be conducted independently of the LCRF-LEADER screening trial, evaluating for efficacy. If none of the 10 oncogenic drivers are detected, the patient will be offered participation in any clinical trial of neoadjuvant therapy available at their treating institution or standard of care therapy. For patients not enrolled on a targeted treatment trial, circulating tumor DNA in blood (ctDNA) will be collected at 3 time points: before neoadjuvant treatment, after neoadjuvant treatment but before surgery, and after surgery. This initiative will be correlated with various clinical outcomes. Prespecified clinical data will be collected for correlation with these circulating biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage IA2-III lung cancers
* Potentially resectable if lung cancer suspicion confirmed pathologically
* Operable

Exclusion Criteria:

* No concurrent malignancy
* No prior lung cancer within last 2 years
* Purely ground glass pulmonary opacity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The LCMC LEADER screening trial will enroll all patients with clinically suspected, resectable stage I-III lung cancers. The population of interest is patients with resectable non-squamous non-small cell lung cancer, however a histologic diagnosis is not required at the time of study enrollment. We anticipate a small portion of patients with squamous cell and non-NSCLC histologies to be genotyped centrally in parallel to their histologic diagnosis. Only patients with non-small cell lung cancers that are not purely squamous will be counted towards the primary study endpoint.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients who Possess Actionable Oncogenic Drivers | 8 weeks
  The primary outcome measure is the determination of the proportion of patients with stage IA2-III lung cancers who possess actionable oncogenic drivers. A patient is considered to have a actionable oncogenic driver if they have any of the following 10 genomic alterations: ALK rearrangements, BRAFV600E mutations, EGFR sensitizing mutations, HER2 mutation, HER2 amplification, MET amplification, MET exon 14 mutation, RET rearrangements, NTRK rearrangement, or ROS1 rearrangements.

SECONDARY OUTCOMES:
Tumor Mutation Burden (TMB) Assessment | 8 weeks
  Measure TMB in all patient tumor samples (Mutations per megabase)

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Swanson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (21):
- United States (21):
  - University of California, Davis, Davis, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - St. Joseph's Hospital Orange, Orange, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - NYU, New York, New York
  - Columbia University, New York, New York
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided